CLINICAL TRIAL: NCT05781828
Title: Noninvasive Methods For Prediction of Esophageal Varices in Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Farag, Resident Doctor, Assiut University
Other Study IDs: Esophageal Varices in Children
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laboratory investigation: Complete blood count, liver function tests, prothrombin time(PT), prothrombin concentration(PC), international normalized ratio (INR), renal chemistry and electrolytes
  Interventions: Diagnostic Test: Detailed abdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Detailed abdominal ultrasound — size of the liver and architecture, size of the spleen, presence or absence of ascites

SUMMARY:
The aim of this study is to use non-invasive methods to identify patients at risk of developing gastrointestinal varices and correlation of these non-invasive methods with the degree of esophageal varices and the presence or absence of risk signs of bleeding such as cherry red spots.

DETAILED DESCRIPTION:
Portal hypertension is the underlying pathophysiological process that leads to the formation of portosystemic collaterals and heralds the onset of a severe complication: variceal hemorrhage. It is estimated that approximately 50% of pediatric patients with chronic liver disease and 90% of those with extrahepatic portal vein obstruction (EHPVO) will experience gastrointestinal bleeding.

Esophagogastroduodenoscopy (EGD) is considered the primary modality for detection and surveillance of esophageal varices (EV) and to determine the risk of bleeding. Varices were graded into four grades I, II, III, and IV according to the Modified Paquet classification. however, invasiveness of the technique and a significant risk associated with sedation on long-term neurological outcomes have limited its use.

Many studies have sought to determine clinical, laboratory, or other noninvasive methods that could predict the presence of EV. Preliminary data suggests that laboratory tests such as platelet count, albumin and ultrasonographic parameters such as presence of splenomegaly, spleen size z score and platelet count to spleen size ratio and the clinical prediction rule (CPR; calculated from platelet count, spleen size z-score, and albumin concentration) may be useful as first-line tools for identification of adults and pediatric patients at risk of variceal development and thus reduce the number of unnecessary EGDs.

ELIGIBILITY:
Inclusion Criteria:

* patients aged < 18 years with a diagnosis of chronic liver disease, extra hepatic portal vein obstruction and/ or liver cirrhosis.

Exclusion Criteria:

* patient who underwent prior variceal treatment (any type) or variceal bleeding prophylaxis (including nonselective β-blocker use, endoscopic variceal ligation or sclerotherapy, surgical portosystemic shunt or transjugular intrahepatic portosystemic shunt insertion), liver transplantation, and malignancy.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients aged < 18 years with a diagnosis of chronic liver disease, extra hepatic portal vein obstruction and/ or liver cirrhosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
noninvasive methods for prediction of esophageal varices in children compared to esophagogastroduodenoscopy results | baseline
  use non-invasive methods to identify patients at risk of developing gastrointestinal varices and correlation of these non-invasive methods with the degree of esophageal varices and the presence or absence of risk signs of bleeding such as cherry red spots.

CONTACTS AND LOCATIONS:
Overall Officials: Emad El-Deen Mahmoud Hammad, Professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt